CLINICAL TRIAL: NCT02629627
Title: Effect of the Administration of Conjugated Linoleic Acid / Leucine Plus Metformin on Visceral Fat in Patients With Metabolic Syndrome
Brief Title: Conjugated Linoleic Acid / Leucine Versus Metformin on Visceral Fat in Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Fernando Grover Paez, Fernando Grover-Paez, PhD, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUCS-INTEC-MV-UKN-001
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Metabolic Syndrome
Keywords: Conjugated Linoleic Acid; Leucine; visceral fat area; Epicardial Fat; Hemodinamic Parameters
MeSH Terms: conditions — Metabolic Syndrome | interventions — Metformin; Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- cojugated ALC/Leucine+Metformin (Experimental): Intervention with conjugated linoleic acid/Leucine + 500mg in individuals with METS
  Interventions: Dietary Supplement: Conjugated linoleic acid/Leucine; Drug: Metformin
- Metformin+placebo conjugatedALC/leucine (Active Comparator): active comparator with Metformin 500mg + Placebo of ACL/Leucine in individuals with METS
  Interventions: Drug: Metformin; Dietary Supplement: Placebo of ACL/Leucine
- Placebo of Metformin (Placebo Comparator): Active comparator with ACL/Leucine + Placebo of Metformin in individuals with METS
  Interventions: Dietary Supplement: Conjugated linoleic acid/Leucine; Other: Placebo of Metformin
- ACL/Leu placebo (Placebo Comparator): Placebo comparator with ACL/Leu placebo + Metformin placebo in individuals with METS
  Interventions: Dietary Supplement: Placebo of ACL/Leucine; Other: Placebo of Metformin

INTERVENTIONS:
Dietary Supplement: Conjugated linoleic acid/Leucine — Conjugated linoleic acid/Leucine capsules, 825mg time daily with the first bite of eat meal during 12 weeks.
  Other Names: UKN
  Arms: Placebo of Metformin; cojugated ALC/Leucine+Metformin
Drug: Metformin — Metformin in a dosis of 500mg per day (with the first bite of the second meal) during 12 weeks
  Other Names: Predial plus
  Arms: Metformin+placebo conjugatedALC/leucine; cojugated ALC/Leucine+Metformin
Dietary Supplement: Placebo of ACL/Leucine — Homologate placebo of ACL/Leucine (linseed oil capsules) in a dosis of 3600 mg each 24 hrs (2 capsules of 2400 mg with the first meal and 1200 mg or 1 capsule with the second meal) during 12 weeks.
  Other Names: Linseed oil
  Arms: ACL/Leu placebo; Metformin+placebo conjugatedALC/leucine
Other: Placebo of Metformin — homologate placebo of metformin (calcinated magnesia) in a dosis of 500 mg per day (with the first bite of the second meal) during 8 weeks
  Other Names: Calcinated magnesia
  Arms: ACL/Leu placebo; Placebo of Metformin

SUMMARY:
In Mexico, obesity is a major public health problem. In recent years he has presented a considerable increase in the population. As a result, it has triggered a proportional increase in the incidence of cardiovascular disease and the development of Metabolic Syndrome (METS). Abdominal obesity is one of the main components of METS which is generally associated with insulin resistance / hyperinsulinemia. This is influenced both by the subcutaneous adipose tissue as visceral adipose tissue. There is evidence that the visceral fat has an important bearing on many factors of METS, like: glucose intolerance, hypertension, dyslipidemia, and insulin resistance.

For management it requires a multidisciplinary approach, including changes in lifestyle, psychological and nutritional intervention as well as pharmacological and non-pharmacological support.

Among non-pharmacological therapies, there is recently the use of Conjugated Linoleic Acid (ACL) and leucine where in its assigned properties include weight reduction, anti-atherogenic , hypocholesterolemic and immunostimulant effect and anticarcinogenic properties. Regarding weight reduction dominates the mechanism of action anti-lipolytic effect. But, studies are needed to link this consumption with the increase or decrease on visceral fat in individuals with METS.

DETAILED DESCRIPTION:
The main objective is to compare the effect of the administration of ACL/Leucine vs. Metformin on visceral fat area in patients with METS. We will conduct a double-blind trial, randomized, on 4 groups, each group with 26 male and female patients of 35-65 years of age with METS diagnosed by IDF criteria. Randomization will determine who will receive the intervention during 8 week trial, each group will be like:

Group (A) intervention with ACL/Leucine plus Metformin: 26 individuals will receive ACL/Leucine in a dosis of 2,475mg per 24 hrs (1,650mg or 2 capsules with the first meal and 825 mg or 1 capsule with the second meal) plus Metformin in a dose of 500 mg per day (with the first bite of the second meal) during 8 weeks.

Group (B) Metformin plus Placebo of ACL/Leucine: 26 individuals will receive Metformin in a dose of 500 mg per day (with the first bite of the second meal) plus homologue placebo of ACL/Leucine (linseed oil capsules) in a dosis of 3600 mg each 24 hrs (2 capsules of 2400 mg with the first meal and 1200 mg or 1 capsule with the second meal) during 8 weeks.

Group (C) ACL/Leucine plus Metformin's Placebo: 26 individuals will receive ACL/Leucine in a dose of 2,475mg per 24 hrs (1,650mg or 2 capsules with the first meal and 825 mg or 1 capsule with the second meal) plus homologate placebo of metformin (calcined magnesia) in a dose of 500 mg per day (with the first bite of the second meal) during 8 weeks.

Group (D) Placebo of ACL/Leucine plus Placebo of Metformin: homologate placebo of ACL/Leucine (linseed oil capsules) in a dose of 3600 mg each 24 hrs (2 capsules of 2400 mg with the first meal and 1200 mg or 1 capsule with the second meal) plus homologated placebo of metformin (calcined magnesia capsules) in a dosis of 500 mg per day (with the first bite of the second meal) during 8 weeks.

The clinical findings and laboratory test include a metabolic profile and biosafety, which will be baseline and at 8 weeks.

Visceral fat area, epicardial fat, body weight, body fat, body mass index (BMI) and blood pressure will be determined during the inicial and final visit, likewise, hemodynamics parameters of arterial stiffness like aortic pulse wave velocity (PWVao), central pulse pressure (PPao), aortic augmentation index (IAxao) and central systolic blood pressure (cSBP) by an oscillometric monitoring system via BPLab ®. Adverse events and adherence to treatment will be documented. Statistical analysis: Mann-Whitney U Test and Wilcoxon exact test. It is considered with significance at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metabolic syndrome by IDF criteria:

  * Central obesity (defi ned as waist circumference* with ethnicity specifi c values)≥80 cm in females and ≥90 cm in males

plus any two of the following four factors:

* Raised triglycerides ≥ 150 mg/dL (1.7 mmol/L) or specific treatment for this lipid abnormality Reduced HDL colesterol
* < 40 mg/dL (1.03 mmol/L) in males < 50 mg/dL (1.29 mmol/L) in females or specifi c treatment for this lipid abnormality
* Raised blood pressure systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg or treatment of previously diagnosed hypertension
* Raised fasting plasma glucose (FPG) ≥ 100 mg/dL (5.6 mmol/L), or previously diagnosed type 2 diabetes

  * Stable body weight in the last 3 months
  * Written informed consent

Exclusion Criteria:

* Ascitis
* With previous abdominal surgery
* Pathologies that course with abdominal wall edema fluid retention
* Paniculitis of reumatic origin or any other ethiology
* Reumatic pathologies
* Metalic prothesis
* Previous known allergy to any of the ingredients that make up the active treatments assigned
* Known problem of fat absortion, esteatorrea, lipase deficiency, malabsortion of intestinal problems, CUCI

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in visceral fat area messure in centimers ^2 at 8 weeks | baseline and 8 weeks
  Before and after intervention using a visceral fat monitor Omron's dual impedance analysis method scan HDS-2000

SECONDARY OUTCOMES:
2. Change from Baseline epicardial fat area messure in milimeters ^2 at 8 weeks | baseline and 8 weeks
  Before and after intervention with ecocardiogragh imagic master of Kontron Medical.
1. Change from Baseline in weight expressed in kg at 8 weeks | baseline and 8 weeks
  Before and after intervention using a tetrapolar bioelectrical impedance analyzer (body composition analyzer TBF-215 - Tanita)
Change from baseline in Body Mass Index, expressed in kg/m^2 at 8 weeks | baseline and 8 weeks
  before and after intervention using a tetrapolar bioelectrical impedance analyzer (body composition analyzer TBF-215 - Tanita)
Change from baseline in Total Tody Fat, expressed in percentage at 8 weeks | baseline and 8 weeks
  before and after intervention using a tetrapolar bioelectrical impedance analyzer (body composition analyzer TBF-215 - Tanita)

OTHER OUTCOMES:
Change from Baseline in central systolic blood pressure in mm/Hg at 8 weeks | baseline and 8 weeks
  Before and after intervention with oscillometric monitoring system via BPLab
Change from Baseline in Pulse Wave Velocity in meters/ second at 8 weeks | baseline and 8 weeks
  Before and after intervention with oscillometric monitoring system via BPLab
Change from Baseline in Fasting plasma glucose in mg/dL at 8 weeks | baseline and 8 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in Total cholesterol in mg/dL at 8 weeks | baseline and 8 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in Triglycerids in mg/dL at 8 weeks | baseline and 8 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in High-density lipoprotein colesterol in mg/dL at 8 weeks | baseline and 8 weeks
  Before and after intervention by friedewall formula
Change from Baseline in Low-density lipoprotein colesterol in mg/dL at 8 weeks | baseline and 8 weeks
  Before and after intervention by friedewall formula
Change from Baseline in Alanine aminotransferase in IU/L at 8 weeks | baseline and 8 weeks
  Before and after intervention by spectrophotometry
Change from Baseline in Aspartate aminotransferase in UI/L at 8 weeks | baseline and 8 weeks
  Before and after intervention by spectrophotometry

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Grover-Páez, PhD, Principal Investigator — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara

IPD SHARING:
Plan to Share IPD: No